CLINICAL TRIAL: NCT03722992
Title: The Effects of Mindfulness-based Stress Reduction on the Urinary Microbiome in Patients With Interstitial Cystitis/Painful Bladder Syndrome
Brief Title: The Effects of Mindfulness-based Stress Reduction in Interstitial Cystitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-056
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2019-11

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Cohort (Other): Mindfulness-based stress reduction (MBSR) treatment group
  Interventions: Other: MBSR

INTERVENTIONS:
Other: MBSR — Guided yoga and meditation practices

SUMMARY:
This is a prospective cohort study to investigate differences in the bladder environment (i.e. urinary microbiome) amongst women with interstitial cystitis (IC) before and after undergoing mindfulness-based stress reduction (MBSR) treatment, including yoga and meditation practices.

DETAILED DESCRIPTION:
Interstitial cystitis (IC), or Painful Bladder Syndrome (PBS) is a debilitating condition of the bladder that is estimated to affect 3-8 million women in the United States. The pathophysiology of the disease is poorly understood, and thus treatment modalities and treatment efficacy vary widely. Lately, much attention has shifted toward investigating how the bladder 'environment' differs amongst women with IC compared to those who do not suffer from IC.

Mindfulness-based stress reduction (MBSR), a complementary alternative medicine (CAM)-based therapy, is a standardized program including components of meditation and yoga. Recent studies show that MBSR improves symptoms in the IC patient population.

The purpose of this study is to compare measurable differences in the urinary microbiome among women with IC before and after MBSR treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* English-speaking
* Established patient of Cincinnati Urogynecology Associates, TriHealth Inc.
* Current diagnosis of IC/PBS, as defined by the American Urological Association (AUA)
* Negative urinalysis or urine culture within 2 months of enrollment
* Currently undergoing first or second-line treatment for IC, as defined by the AUA
* Willingness to participate in study

Exclusion Criteria:

* Non-English speaking
* Unwillingness to participate in study
* Pregnancy or breastfeeding
* Physical or mental impairment that would affect the subject's ability to participate in the MBSR treatment, including patients with Dementia, Parkinsonism, or those who have impaired mobility or hearing
* Current or expected prolonged catheterization
* Expected travel or surgery that would hinder the ability to attend all eight MBSR sessions
* Undergoing third-, fourth-, fifth-, or sixth-line treatment for IC as defined by the AUA
* Subjects on antibiotics currently or prior use within one week of consenting

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Difference in the urinary microbiome before and after MBSR treatment | Before intervention and after completion of the intervention, up to 9 weeks
  Urinary microbiome sequencing analysis will be performed by Resphera Biosciences Laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- TriHealth - Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No